CLINICAL TRIAL: NCT01889238
Title: A PHASE 2, SINGLE-ARM, OPEN-LABEL, MULTICENTER STUDY OF THE CLINICAL ACTIVITY AND SAFETY OF ENZALUTAMIDE IN PATIENTS WITH ADVANCED, ANDROGEN RECEPTOR-POSITIVE, TRIPLE-NEGATIVE BREAST CANCER
Brief Title: Safety and Efficacy Study of Enzalutamide in Patients With Advanced, Androgen Receptor-Positive, Triple Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Astellas Pharma Inc (Industry); Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDV3100-11; 2013-000698-57 (EudraCT Number); C3431007 (Other: Alias Study Number)
Record Dates: First submitted 2013-06-26; First posted 2013-06-28 (Estimated); Results first posted 2018-08-22 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-11

CONDITIONS: Advanced, Androgen Receptor Positive Triple Negative Breast Cancer
Keywords: breast cancer; triple negative; androgen receptor positive
MeSH Terms: conditions — Breast Neoplasms | interventions — enzalutamide

ARMS (1):
- Enzalutamide (Experimental): 160 mg administered as four 40 mg soft gelatin capsules orally once daily
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — 160 mg administered as four soft gelatin capsules orally once daily
  Other Names: Xtandi®; MDV3100

SUMMARY:
The purpose of this study is to determine if enzalutamide is safe and effective in the treatment of patients with advanced breast cancer that express the androgen receptor but do not express the estrogen or progesterone receptor and are not Her2 amplified.

ELIGIBILITY:
Inclusion Criteria:

* Women at least 18 years of age;
* Advanced AR+ TNBC;
* Availability of a representative tumor specimen:
* Either measurable disease or bone only nonmeasurable disease;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.

Exclusion Criteria:

* Any severe concurrent disease, infection, or comorbid condition;
* Any condition or reason that interferes with the patient's ability to participate in the trial, that may cause undue risk, or complicates the interpretation of safety data;
* Current or previously treated brain metastasis or active leptomeningeal disease;
* Current hormone replacement therapy;
* Local palliative radiation therapy within 7 days before day 1;
* History of another invasive cancer within 5 years of day 1;
* Absolute neutrophil count < 1500/µL, platelet count < 75,000/µL, or hemoglobin < 9 g/dL (5.6 mmol/L) at the screening visit;
* Creatinine > 1.5 times upper limit of normal (ULN) at the screening visit;
* History of seizure or any condition that may predispose to seizure;
* Clinically significant cardiovascular disease;
* Active gastrointestinal disorder affecting absorption;
* Major surgery within 4 weeks before day 1;
* Treatment with any commercially available anticancer agent within 14 days before day 1;
* Treatment with any investigational agent within 2 weeks before day 1;
* Treatment with any of the following medications within 2 weeks before day 1: Estrogens, including hormone replacement therapy; Androgens (testosterone, dihydroepiandrosterone, etc);Systemic radionuclides (eg, samarium or strontium);Vaccine therapy;
* Hypoglycemic episode requiring medical intervention while on insulin treatment within 12 months before day 1;
* Hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 118 (Actual)
Dates: Start 2013-06-12 (Actual); Primary Completion 2015-03-01 (Actual); Study Completion 2024-01-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer; Pfizer CT.gov Call Center, Study Chair — Pfizer
Locations (116):
- United States (81):
  - Rocky Mountain Cancer Centers, Colorado Springs, Colorado
  - Rocky Mountain Cancer Centers, Lakewood, Colorado
  - Rocky Mountain Cancer Center Sky Ridge, Lone Tree, Colorado
  - Rocky Mountain Cancer Centers, Lone Tree, Colorado
  - Florida Cancer Specialists, Altamonte Springs, Florida
  - Florida Cancer Specialists, Bonita Springs, Florida
  - Florida Cancer Specialists, Bradenton, Florida
  - Florida Cancer Specialists, Brandon, Florida
  - Florida Cancer Specialists, Cape Coral, Florida
  - Florida Cancer Specialists, Clearwater, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Florida Cancer Specialist South Division, Fort Myers, Florida
  - Florida Cancer Specialists, Gainesville, Florida
  - Florida Cancer Specialists, Hudson, Florida
  - Florida Cancer Specialists, Largo, Florida
  - Florida Cancer Specialists, Naples, Florida
  - Florida Cancer Specialists, New Port Richey, Florida
  - Florida Cancer Specialists, Orange City, Florida
  - Florida Cancer Specialists, Orlando, Florida
  - Florida Cancer Specialists, Port Charlotte, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Florida Cancer Specialists, Spring Hill, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Florida Cancer Specialists, Tampa, Florida
  - Florida Cancer Specialists, Tavares, Florida
  - Florida Cancer Specialists, Venice, Florida
  - Northwestern Medical Faculty Foundation(NMFF)/ Women's Cancer Center Shared Laboratories, Chicago, Illinois
  - Northwestern Medical Faculty Foundation, Chicago, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - The University of Chicago Medical Center, Investigational Drug Service Department of Pharmacy, Chicago, Illinois
  - The University of Chicago, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center at Silver Cross Hospital, New Lenox, Illinois
  - Indiana University Health Hospital, Indianapolis, Indiana
  - Indiana University Health Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Investigational Drug Services, Indianapolis, Indiana
  - Sidney and Lois Eskenazi Hospital, Indianapolis, Indiana
  - Springmill Medical Clinic, Indianapolis, Indiana
  - Oncology Hematology Care, Inc., Crestview Hills, Kentucky
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - The West Clinic, PC, Corinth, Mississippi
  - The West Clinic, PC, Southaven, Mississippi
  - Siteman Cancer Center, City of Saint Peters, Missouri
  - Barnes-Jewish Hospital, St Louis, Missouri
  - Washington University Infusion Center Pharmacy, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center-West County, St Louis, Missouri
  - Hematology Oncology Associates of Northern NJ, Morristown, New Jersey
  - Memorial Sloan Kettering - I Chemotherapy Practice/Investigational Drug Service, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Cone Health Cancer Center, Greensboro, North Carolina
  - Wesley Long Community Hospital, Greensboro, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Oncology Hematology Care, Inc., Fairfield, Ohio
  - Greenville Health System, Greenville, South Carolina
  - Greenville Health System, Seneca, South Carolina
  - Greenville Health System, Spartanburg, South Carolina
  - Tennessee Oncology, PLLC, Dickson, Tennessee
  - Tennessee Oncology, PLLC, Franklin, Tennessee
  - Tennessee Oncology, PLLC, Gallatin, Tennessee
  - Tennessee Oncology, PLLC, Hermitage, Tennessee
  - Tennessee Oncology, PLLC, Lebanon, Tennessee
  - The West Clinic, PC, Memphis, Tennessee
  - Tennessee Oncology, PLLC, Murfreesboro, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - The Sarah Cannon Research Institute, Nashville, Tennessee
  - Vanderbilt Breast Center at One Hundred Oaks, Nashville, Tennessee
  - Vanderbilt Health Pharmacy One Hundred Oaks, Nashville, Tennessee
  - Henry-Joyce Cancer Clinic, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Smyrna, Tennessee
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - Texas Oncology - Memorial City, Houston, Texas
  - Texas Oncology - Longview Cancer Center, Longview, Texas
  - Texas Oncology-Tyler, Tyler, Texas
  - Virginia Cancer Institute, Mechanicsville, Virginia
  - Virginia Cancer Institute, Midlothian, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Oncology Associates, Norfolk, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Virginia Oncology Associates, Virginia Beach, Virginia
- Belgium (2):
  - UZA, Edegem, Antwerpen
  - Institut Jules Bordet, Brussels
- Canada (3):
  - British Columbia Cancer Agency - Vancouver Centre, Vancouver, British Columbia
  - Sunnybrook Research Institute, Toronto, Ontario
  - McGill University Health Centre-Cedars Cancer Centre, Montreal, Quebec
- Ireland (9):
  - Department of Radiology, Dooradoyle, Limerick
  - 3rd Floor,Oncology Link office, Dublin
  - Department of Radiology, Dublin
  - Institute for Cancer Research, Dublin
  - Mater Private Hospital, Dublin
  - Pharmacy Department, Dublin
  - Radiology Department, Dublin
  - Cancer Clinical Trials Unit, Mid-Western Cancer center, Limerick
  - Pharmacy Department, Limerick
- Italy (4):
  - Dipartimento di Oncologia Medica, IRCCS Ospedale San Raffaele, Milan
  - Farmacia (magazzino ricevimento merc), IRCCS Ospedale San Raffaele, Milan
  - U.O Farmaceutica, Nuovo Ospedale di Prato Palazzina dei servizi, Prato
  - U.O. Oncologia Medica, Nuovo Ospedale di Prato, Prato
- Spain (7):
  - Hospital Universitario HM Monteprincipe, Boadilla del Monte, Madrid
  - Grupo Hospitalario Quiron - Hospital Quiron Barcelona, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon Y Cajal, Madrid
  - Hospital Universitario 12 Octubre, Madrid
  - Centro Intergral Oncologico Clara Campal, Madrid
  - Hospital de Madrid Norte-Sanchinarro., Madrid
- United Kingdom (10):
  - Clinical Investigation and Research Unit, Brighton, England
  - Pharmacy Department, Brighton, England
  - Radiation Safety Service, Medical Physics Department, Brighton, England
  - Histopathology Department, Nottingham, England
  - Nottingham University Hospital, Nottingham, England
  - Pharmacy Department, Nottingham, England
  - Radiology Department, Nottingham, England
  - Department of Radiology, Truro, England
  - Pharmacy Department, Truro, England
  - Royal Cornwall Hospitals NHS trust, Truro, Cornwall, England

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Kumar V, Yu J, Phan V, Tudor IC, Peterson A, Uppal H. Androgen Receptor Immunohistochemistry as a Companion Diagnostic Approach to Predict Clinical Response to Enzalutamide in Triple-Negative Breast Cancer. JCO Precis Oncol. 2017 Nov;1:1-19. doi: 10.1200/PO.17.00075. PMID 35172518
- [Derived] Traina TA, Miller K, Yardley DA, Eakle J, Schwartzberg LS, O'Shaughnessy J, Gradishar W, Schmid P, Winer E, Kelly C, Nanda R, Gucalp A, Awada A, Garcia-Estevez L, Trudeau ME, Steinberg J, Uppal H, Tudor IC, Peterson A, Cortes J. Enzalutamide for the Treatment of Androgen Receptor-Expressing Triple-Negative Breast Cancer. J Clin Oncol. 2018 Mar 20;36(9):884-890. doi: 10.1200/JCO.2016.71.3495. Epub 2018 Jan 26. PMID 29373071

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Total of 118 participants with advanced androgen receptor positive (AR+) and triple-negative breast cancer (TNBC) were enrolled at total of 34 study sites in North America and Europe to attain total of 78 evaluable participants.
Groups:
- Enzalutamide: Participants received enzalutamide 160 mg (as four 40 mg soft gelatin capsules), orally once daily until disease progression, intolerable AEs (including any seizures), non-compliance with protocol requirements, initiation of a new anti-tumor treatment, or participant or physician decision to discontinue treatment or death due to any cause.
Period: Overall Study
Arm/Group | Enzalutamide
Started | 118
Completed | 0
Not Completed | 118
Not completed — Death | 1
Not completed — Withdrawal by Subject | 1
Not completed — Adverse Event | 6
Not completed — Disease Progression | 104
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all enrolled participants who had positive androgen receptor (AR+) breast cancer as assessed by central review and received at least 1 dose of study drug.
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.3 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 108
  Unknown or Not Reported | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 91
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Clinical Benefit at Week 16: Evaluable Population
Description: Percentage of participants with a clinical benefit at Week 16 defined as percentage of participants with a best response of complete response (CR), partial response(PR), stable disease(SD) for >=16 weeks on radiologic imaging based on Investigator assessment using Response Evaluation Criteria in Solid Tumors version 1.1(RECIST 1.1). An estimate of the percentage and its exact 2-sided 85% confidence interval(CI) were calculated using the Blaker method. As per RECIST 1.1, CR defined as disappearance of all target, non-target lesions and normalization of tumor marker level and all lymph nodes decreased to non-pathological in size <10mm short axis. PR: At least 30% decrease in sum of longest diameter (LD) of target lesions taking as reference baseline sum of LD, without progression of non-target lesions, no appearance of new lesions. SD: Neither sufficient reduction to qualify as PR nor sufficient increase to qualify as PD, using the smallest sum diameters during the study as a reference.
Time Frame: Week 16
Population: Evaluable population included all enrolled participants who had centrally assessed AR + breast cancer (total nuclear AR expression in >= 10% of tumor cells), had at least 1 dose of study drug and had at least 1 available post baseline tumor assessment evaluable as per RECIST 1.1.
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 78
Percentage of participants | 33.3 [25.53 to 41.63]

2. Primary Outcome: Percentage of Participants With Clinical Benefit at Week 16: Intent-to-Treat (ITT) Population
Description: Percentage of participants with a clinical benefit at Week 16 defined as percentage of participants with a best response of CR, PR, or SD for >= 16 weeks on radiologic imaging based on Investigator assessment using RECIST 1.1. An estimate of the percentage and its exact 2-sided 85% CI were calculated using the Blaker method. As per RECIST 1.1, CR defined as disappearance of all target, non-target lesions and normalization of tumor marker level and all lymph nodes decreased to non-pathological in size <10 mm short axis. PR: At least 30% decrease in sum of LD of target lesions taking as reference baseline sum of LD, without progression of non-target lesions, no appearance of new lesions. SD: Neither sufficient reduction to qualify as PR nor sufficient increase to qualify as PD, using the smallest sum diameters during the study as a reference.
Time Frame: Week 16
Population: ITT population included all enrolled participants who had centrally assessed AR+ breast cancer and received at least 1 dose of study drug.
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Percentage of participants | 24.6 [18.98 to 30.88]

3. Secondary Outcome: Percentage of Participants With Clinical Benefit at Week 24: Evaluable Population
Description: Percentage of participants with a clinical benefit at Week 24 defined as percentage of participants with a best response of CR, PR, or SD for >= 24 weeks on radiologic imaging based on investigator assessment using RECIST 1.1. An estimate of the percentage and its exact 2-sided 85% CI were calculated using the Blaker method. As per RECIST 1.1, CR defined as disappearance of all target, non-target lesions and normalization of tumor marker level and all lymph nodes decreased to non-pathological in size <10 mm short axis. PR: At least 30% decrease in sum of LD of target lesions taking as reference baseline sum of LD, without progression of non-target lesions, no appearance of new lesions. SD: Neither sufficient reduction to qualify as PR nor sufficient increase to qualify as PD, using the smallest sum diameters during the study as a reference.
Time Frame: Week 24
Population: as for outcome 1
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 78
Percentage of participants | 28.2 [21.04 to 36.48]

4. Secondary Outcome: Percentage of Participants With Clinical Benefit at Week 24: ITT Population
Description: as for outcome 3
Time Frame: Week 24
Population: as for outcome 2
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Percentage of participants | 20.3 [15.16 to 26.21]

5. Secondary Outcome: Percentage of Participants With Best Objective Response: Evaluable Population
Description: Percentage of participants with best objective response defined as percentage of participants with a best response of CR and PR based on investigator assessment of target, non-target and new lesions using RECIST 1.1. As per RECIST 1.1, CR defined as disappearance of all target, non-target lesions and normalization of tumor marker level and all lymph nodes decreased to non-pathological in <10 mm short axis. PR: At least 30% decrease in sum of LD of target lesions taking as reference baseline sum of LD, without progression of non-target lesions, no appearance of new lesions.
Time Frame: From Baseline up to disease progression or death due to any cause (up to 87 Weeks)
Population: Evaluable population included all enrolled participants who had centrally assessed AR + breast cancer (total nuclear AR expression in >= 10% of tumor cells), had at least 1 dose of study drug and had at least 1 available post baseline tumor assessment evaluable as per RECIST 1.1. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Percentage of participants | 8.5 [3.05 to 12.02]

6. Secondary Outcome: Percentage of Participants With Best Objective Response: ITT Population
Description: as for outcome 5
Time Frame: From Baseline up to disease progression or death due to any cause (up to 87 Weeks)
Population: ITT population included all enrolled participants who had centrally assessed AR+ breast cancer and received at least 1 dose of study drug. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Number (85% Confidence Interval); unit: Percentage of participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 97
Percentage of participants | 6.2 [2.80 to 8.95]

7. Secondary Outcome: Progression-Free Survival (PFS): Evaluable Population
Description: PFS was defined as the time (in weeks) from the date of first dose of study drug to the date of documented disease progression or death due to any cause whichever occurs first as determined by the investigator using RECIST 1.1. As per RECIST 1.1, progression was defined as: >=20 percent increase in sum of LD of target lesions taking as a reference the smallest sum of the LD recorded since the treatment started, or the appearance of one or more new lesions and/or unequivocal progression of existing non target-lesions.
Time Frame: From Baseline up to disease progression or death due to any cause (up to 87 Weeks)
Population: as for outcome 5
Measure: Median (85% Confidence Interval); unit: Weeks
Arm/Group | Enzalutamide
Number analyzed (Participants) | 78
Weeks | 14.3 [8.3 to 16.1]

8. Secondary Outcome: Progression-Free Survival: ITT Population
Description: as for outcome 7
Time Frame: From Baseline up to disease progression or death due to any cause (up to 87 Weeks)
Population: as for outcome 2
Measure: Median (85% Confidence Interval); unit: Weeks
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Weeks | 12.6 [8.1 to 15.1]

9. Other Pre Specified Outcome: Trough Plasma Concentration of Enzalutamide and Its Metabolite
Description: M2 was the metabolite of enzalutamide. The lower limit of quantitation (LLQ) was 0.0200 micrograms per milliliter (mcg/mL) for enzalutamide and M2.
Time Frame: Predose on Day 1 (Baseline), Week 9 and Week 17
Population: Pharmacokinetics (PK) analysis population included all participants who received 1 dose or partial dose of study drug, and who had at least 1 enzalutamide or M2 plasma concentration assessment. Here, 'Number of Participants Analyzed' signifies participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mcg/mL
Arm/Group | Enzalutamide
Number analyzed (Participants) | 115
mcg/mL
  Enzalutamide: Day 1 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol, values below the limit of quantitation (BLQ) were set to missing and hence not reported.
  M2: Day 1 | NA (NA) — None of the participants had data above LLQ and as per the predefined protocol, values below the limit of quantitation (BLQ) were set to missing and hence not reported.
  Enzalutamide: Week 9 | 12.59 (33.46)
  M2: Week 9 | 13.48 (35.64)
  Enzalutamide: Week 17 | 12.79 (37.33)
  M2: Week 17 | 13.88 (25.47)

10. Other Pre Specified Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment emergent are events that were absent before treatment or that worsened relative to pretreatment state between first dose of study drug and up to 30 days after last dose of study drug or the day prior to initiation of new anti-tumor treatment. AEs included both serious and non-serious AEs.
Time Frame: Baseline up to 87 weeks
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants
  Treatment emergent adverse events | 109
  Treatment emergent serious adverse events | 29

11. Other Pre Specified Outcome: Number of Participants With Study Drug Discontinuation Due to Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Data reported here is for study drug discontinuation due to adverse events.
Time Frame: Baseline up to 87 weeks
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants | 8

12. Other Pre Specified Outcome: Number of Participants With Grade 3 or Higher Adverse Events
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Severity of the AEs was graded according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. As per the NCI CTCAE, version 4.0, Grade 3= severe, Grade 4= life-threatening and Grade 5= death. Only the participants with treatment-emergent AEs of Grade 3 (severe) or higher grade were reported in this outcome measure.
Time Frame: Baseline up to 87 weeks
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants | 36

13. Other Pre Specified Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Criteria: Systolic blood pressure (SBP):absolute SBP<90 millimeters of mercury (mmHg) and decrease from baseline (DFB)>30mmHg, absolute SBP>180mmHg and increase from baseline (IFB)>40 mmHg, final visit (FV) or 2 consecutive visits (CV) SBP>=20 mmHg change from baseline (CFB), most extreme post-baseline SBP>=140mmHg, most extreme post- baseline SBP>=180mmHg, most extreme SBP>=140mmHg and>=20 mmHg CFB, most extreme SBP>=180mmHg and>=20mmHg CFB; diastolic blood pressure (DBP): absolute DBP>105mmHg and IFB>30mmHg, absolute DBP<50mmHg and DFB>20mmHg, final visit or 2 consecutive visits DBP>=15mmHg CFB, most extreme post-baseline DBP>=90mmHg, most extreme post-baseline DBP>=105mmHg, most extreme DBP>=90mmHg and>=15mmHg CFB, most extreme DBP>=105mmHg and>=15mmHg CFB; heart rate<50beats per minute (BPM) and DFB>20BPM or heart rate>120BPM and IFB>30BPM. Only those categories, in which at least 1 participant had data were reported.
Time Frame: From start of study treatment on Day 1 up to 30 days after the last dose of study drug (up to maximum of 9.6 years)
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants
  SBP:Most extreme SBP>=140 mmHg and>=20 mmHg CFB | 12
  SBP: absolute SBP <90 mmHg and DFB>30 mmHg | 1
  SBP: Most extreme post baseline SBP >=140 mmHg | 42
  SBP: Most extreme post baseline SBP >=180 mmHg | 1
  DBP:Most extreme DBP>=90 mmHg and>=15 mmHg CFB | 12
  DBP:Most extreme DBP>=105 mmHg and>=15 mmHg CFB | 2
  DBP: Most extreme post baseline result >=90 mmHg | 24
  DBP: Most extreme post baseline result >=105 mmHg | 4

14. Other Pre Specified Outcome: Number of Participants With Change From Baseline in Laboratory Parameters Grades by 2 or More Grades
Description: Laboratory tests included hematology parameters [low lymphocytes (10^6/L), white blood cells (10^9/L), neutrophils (10^6/L), hemoglobin gram per Liter(g/L) and platelets (10^9/L)] and chemistry parameters [mean albumin grams per Liter(g/L), calcium milli mole per Liter(mmol/L), Phosphate (mmol/L), alanine aminotransferase units per Liter(U/L), Aspartate aminotransferase (U/L), bilirubin micro mole per Liter, Alkaline phosphatase (U/L) and glucose (mmol/L)]. Number of participants with change from baseline in laboratory parameters Grades by 2 or More Grades as per NCI-CTCAE (version 4.0) (Grade 2=Moderate, Grade 3= Severe, Grade 4= Life-threatening) were reported.
Time Frame: From start of study treatment on Day 1 up to 30 days after the last dose of study drug (up to maximum of 9.6 years)
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants
  Hematology: Hemoglobin | 1
  Hematology: Leukocytes | 4
  Hematology: Lymphocytes | 12
  Hematology: Neutrophils | 2
  Hematology: Platelets | 1
  Chemistry: Alanine aminotransferase | 1
  Chemistry: Albumin | 4
  Chemistry: Alkaline phosphatase | 5
  Chemistry: Bilirubin | 2
  Chemistry: Calcium | 2
  Chemistry: Glucose | 5
  Chemistry: Phosphate | 4
  Chemistry: Aspartate Aminotransferase | 1

15. Secondary Outcome: Time to Response: Evaluable Population
Description: The time to response is defined as the time from the date of first dose of study drug to initial CR or PR. Participants without response of CR or PR before the data cutoff date were censored at the last tumor assessment date before the data cutoff. Kaplan-Meier method was used to summarize time to response.
Time Frame: From first dose of study drug until first documentation of CR or PR or data censoring date, whichever occurred first (up to 87 Weeks)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Weeks | NA [NA to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with the event.

16. Secondary Outcome: Duration of Response: Evaluable Population
Description: Duration of objective response is defined as the time from initial CR or PR to documented disease progression or death due to any cause, whichever occurs first. Participants without disease progression or death due to any cause before the data cutoff date were censored at the last tumor assessment date before the data cutoff.
Time Frame: From first documentation of CR or PR until first documentation of tumor progression or death due to any cause or data censoring date, whichever occurred first (up to 87 Weeks)
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | Enzalutamide
Number analyzed (Participants) | 59
Weeks | NA [NA to NA] — Median and 95%CI could not be estimated due to insufficient number of participants with the event.

17. Secondary Outcome: Number of Participants With Postbaseline Laboratory Toxicities Grade 3 or 4
Description: Laboratory parameters included hematology parameters [low lymphocytes (10^6/L), neutrophils (10^6/L) and Leukocytes (10^9/L)] and chemistry parameters [high phosphate (mmol/L), bilirubin, Alkaline phosphatase (U/L) and glucose (mmol/L)]. Number of participants with postbaseline laboratory toxicity Grade 3 or 4 as per NCI-CTCAE (version 4.0) (Grade 3= Severe, Grade 4= Life-threatening) were reported.
Time Frame: From start of study treatment on Day 1 up to 30 days after the last dose of study drug (up to maximum of 9.6 years)
Population: Safety population included all participants who received 1 dose or partial dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Enzalutamide
Number analyzed (Participants) | 118
Participants
  Hematology: Leukocytes | 1
  Hematology: Lymphocytes | 9
  Hematology: Neutrophils | 1
  Chemistry: Alkaline Phosphatase | 1
  Chemistry: Bilirubin | 1
  Chemistry: Glucose | 4
  Chemistry: Phosphate | 1

ADVERSE EVENTS:
Time Frame: Baseline up to 87 weeks
Description: Same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. AEs and SAEs were collected for safety population.
Arm/Group | Enzalutamide
All-Cause Mortality (participants affected / at risk) | 88/118
Serious Adverse Events (participants affected / at risk) | 29/118
Other Adverse Events (participants affected / at risk) | 106/118
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=118)
Pericardial effusion (Cardiac disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Disease progression (General disorders) | 3
General physical health deterioration (General disorders) | 1
Pain (General disorders) | 1
Bile duct obstruction (Hepatobiliary disorders) | 1
Lung infection (Infections and infestations) | 2
Sepsis (Infections and infestations) | 2
Cellulitis (Infections and infestations) | 1
Device related infection (Infections and infestations) | 1
Respiratory tract infection (Infections and infestations) | 1
Soft tissue infection (Infections and infestations) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Radiation oesophagitis (Injury, poisoning and procedural complications) | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1
Traumatic fracture (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Breast cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Spinal cord compression (Nervous system disorders) | 2
Cognitive disorder (Nervous system disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Enzalutamide (N=118)
Nausea (Gastrointestinal disorders) | 40
Fatigue (General disorders) | 49
Diarrhoea (Gastrointestinal disorders) | 18
Constipation (Gastrointestinal disorders) | 17
Vomiting (Gastrointestinal disorders) | 11
Abdominal pain (Gastrointestinal disorders) | 7
Pain (General disorders) | 9
Asthenia (General disorders) | 6
Nasopharyngitis (Infections and infestations) | 6
Weight decreased (Investigations) | 8
Decreased appetite (Metabolism and nutrition disorders) | 22
Back pain (Musculoskeletal and connective tissue disorders) | 17
Arthralgia (Musculoskeletal and connective tissue disorders) | 18
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Headache (Nervous system disorders) | 17
Dizziness (Nervous system disorders) | 6
Neuropathy peripheral (Nervous system disorders) | 6
Insomnia (Psychiatric disorders) | 17
Anxiety (Psychiatric disorders) | 7
Breast pain (Reproductive system and breast disorders) | 6
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Cough (Respiratory, thoracic and mediastinal disorders) | 8
Hot flush (Vascular disorders) | 12
Upper respiratory tract infection (Infections and infestations) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.